CLINICAL TRIAL: NCT01231971
Title: Alzheimer's Disease Neuroimaging Initiative 2
Acronym: ADNI2
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Northern California Institute of Research and Education (Other); National Institute on Aging (NIA) (NIH); Alzheimer's Therapeutic Research Institute (Other)
Responsible Party: Principal Investigator, Paul S. Aisen, Professor, University of Southern California
Other Study IDs: ADC-039-ADNI2; U01AG024904 (NIH)
Record Dates: First submitted 2010-10-27; First posted 2010-11-01 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment (MCI); Alzheimer's Disease (AD); Significant Memory Concern (SMC); Early Mild Cognitive Impairment (EMCI); Late Mild Cognitive Impairment (LMCI)
Keywords: amyloid; plaques; neuroimaging; biomarkers; cognition disorder; early detection; Amnestic MCI; pre-dementia; dementia; Alzheimer's disease; tau
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Plaque, Amyloid; Cognition Disorders; Dementia; Pick Disease of the Brain | interventions — florbetapir; 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (5):
- Cognitively Normal (CN): 150 newly enrolled participants with no apparent memory problems, and CN participants followed from the ADNI1 study
  Interventions: Drug: Florbetapir; Drug: Flortaucipir
- Early Mild Cognitive Impairment (EMCI): 100 newly enrolled early amnestic MCI participants, and approximately 200 EMCI participants will be followed from the ADNI-GO study
  Interventions: Drug: Florbetapir; Drug: Flortaucipir
- Late Mild Cognitive Impairment (LMCI): 150 newly enrolled late MCI participants, and LMCI participants followed from the ADNI1 study
  Interventions: Drug: Florbetapir; Drug: Flortaucipir
- Alzheimer's Disease (AD): 150 newly enrolled mild AD participants
  Interventions: Drug: Florbetapir; Drug: Flortaucipir
- Significant Memory Concern (SMC): 100 newly enrolled participants with Significant Memory Concern (SMC)
  Interventions: Drug: Florbetapir; Drug: Flortaucipir

INTERVENTIONS:
Drug: Florbetapir — Participants will receive a single bolus intravenous injection of 10 mCi (370 MBq) (+/- 10%) florbetapir F18. At approximately 50-minutes post dose, scanning will begin. An approximately 20-minute image acquisition scan will be performed.
  Other Names: 18F-AV-45, LY3078786
Drug: Flortaucipir — Participants will receive a single bolus intravenous injection of 10 mCi (370 MBq) flortaucipir injection followed by a saline flush. At approximately 75-minutes post dose, scanning will begin. An approximately 30-minute image acquisition scan will be performed.
  Other Names: 18F-AV-1451 (also known as [F-18]T807 or LY3191748)

SUMMARY:
The purpose of this study is to build upon the information obtained in the original Alzheimer's Disease Neuroimaging Initiative (ADNI1) and ADNI-GO (Grand Opportunity; a study funded through an NIH grant under the American Recovery and Reinvestment Act), to examine how brain imaging technology can be used with other tests to measure the progression of mild cognitive impairment (MCI) and early Alzheimer's disease (AD). ADNI2 seeks to inform the neuroscience of AD. This information will aid in the early detection of AD, and in measuring the effectiveness of treatments in future clinical trials.

DETAILED DESCRIPTION:
The Alzheimer's Disease Neuroimaging Initiative (ADNI) began in October 2004 as a landmark study with a public-private partnership that gathered and analyzed thousands of brain scans, genetic profiles and biomarkers in blood and cerebrospinal fluid (CSF). Although the original goal was to define biomarkers for use in clinical trials to determine the best way to measure treatment effects of Alzheimer's disease (AD), the goal has been expanded to using biomarkers to identify AD at a pre-dementia stage. ADNI1 involves scientists at 59 research centers, 54 in the U.S. and five in Canada. Originally 800 participants were enrolled. This group was comprised of 200 participants with AD, 400 with mild cognitive impairment (MCI) and 200 with normal cognition. In ADNI-GO, an estimated 200 participants with early amnestic MCI (EMCI) were enrolled to understand and characterize the mildest symptomatic phase of AD. An additional 650 participants will be enrolled under ADNI2.

Some of the leading-edge technologies under study are brain-imaging techniques, such as positron emission tomography (PET), including FDG-PET (which measures glucose metabolism in the brain); PET using a radioactive compound (Florbetapir F 18) that measures brain beta-amyloid; and structural MRI. Brain scans are showing scientists how the brain's structure and function change as AD starts and progresses. Biomarkers in cerebrospinal fluid are revealing other changes that could identify which patients with MCI will develop Alzheimer's. Scientists are looking at levels of beta-amyloid and tau in cerebrospinal fluid. (Abnormal amounts of the amyloid and tau proteins in the brain are hallmarks of Alzheimer's disease.)

ADNI2 extends the work of ADNI1 and ADNI GO to understand the progression of AD. The overall goal is to determine the relationships among the clinical, cognitive, imaging, genetic and biochemical biomarker characteristics of the entire spectrum of AD, as the pathology evolves from normal aging through very mild symptoms, to MCI, to dementia.

The overall impact of this study will be increased knowledge concerning the sequence and timing of events leading to MCI and AD, development of better clinical and imaging/fluid biomarker methods for early detection and for monitoring the progression of these conditions, and facilitation of clinical trials to slow disease progression, ultimately contributing to the prevention of AD.

ELIGIBILITY:
Inclusion Criteria:

Participants will be classified as either normal controls, SMC, EMCI, LMCI or AD participants. General Inclusion Criteria will apply to all groups, with specific criteria for each group as described below:

General (applies to each category):

* Geriatric Depression Scale less than 6.
* Age between *55-90 (inclusive). *For normal controls and SMC participants, age must be between 65-90.
* Study partner is available who has frequent contact with the participant (e.g. an average of 10 hours per week or more), and can accompany the participant to all clinic visits for the duration of the protocol.
* Visual and auditory acuity adequate for neuropsychological testing.
* Good general health with no diseases expected to interfere with the study.
* Participant is not pregnant, lactating, or of childbearing potential (i.e. women must be two years post-menopausal or surgically sterile).
* Willing and able to participate in a longitudinal imaging study.
* Hachinski less than or equal to 4.
* Completed six grades of education or has a good work history (sufficient to exclude mental retardation).
* Must speak English or Spanish fluently.
* Willing to undergo repeated MRIs (3Tesla) and at least two PET scans (one FDG and one Amyloid imaging) and no medical contraindications to MRI.
* Agrees to collection of blood for Genome Wide Association Studies (GWAS), APOE testing and DNA and RNA banking.
* Agrees to collection of blood for biomarker testing.
* Agrees to at least one lumbar puncture for the collection of CSF.

Specific Inclusion Criteria for normal controls:

* Participant must be free of memory complaints, verified by a study partner.
* Normal memory function score on Wechsler Memory Scale (adjusted for education)
* Mini-Mental State Exam (MMSE) score between 24 and 30 (inclusive)
* Clinical Dementia Rating (CDR) = 0; Memory Box score must be 0
* Cognitively normal, based on an absence of significant impairment in cognitive functions or activities of daily living
* Stability of Permitted Medications for 4 weeks. In particular, participants may take:

  * Antidepressants lacking significant anticholinergic side effects
  * Estrogen replacement therapy is permissible
  * Gingko biloba is permissible, but discouraged
  * Washout from psychoactive medication (e.g., excluded antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics, etc.) for at least 4 weeks prior to screening

Specific Inclusion Criteria for SMC participants:

* Subjects that are "self-referrals" that have a significant subjective memory concern
* Significant memory concern confirmed by a Cognitive Change Index score of more than or equal to 16
* Normal memory function score on Wechsler Memory Scale (adjusted for education)
* Mini-Mental State Exam (MMSE) score between 24 and 30 (inclusive)
* Clinical Dementia Rating (CDR) = 0; Memory Box score must be 0
* Cognitively normal, based on the absence of significant memory impairment in cognitive function or activities of daily living
* Stability of Permitted Medications for 4 weeks. In particular, subjects may take:

  * Antidepressants lacking significant anticholinergic side effects
  * Estrogen replacement therapy is permissible
  * Gingko biloba is permissible, but discouraged
  * Washout from psychoactive medication (e.g., excluded antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics, etc.) for at least 4 weeks prior to screening

Specific Inclusion Criteria for EMCI and LMCI participants:

* Participant must have a subjective memory concern as reported by participant, study partner, or clinician
* Abnormal memory function score on Wechsler Memory Scale (adjusted for education)
* Mini-Mental State Exam (MMSE) score between 24 and 30 (inclusive)
* Clinical Dementia Rating (CDR) = 0.5; Memory Box score must be at least 0.5
* General cognition and functional performance sufficiently preserved such that a diagnosis of AD cannot be made by the site physician at the time of the screening visit
* Stability of Permitted Medications for 4 weeks. In particular, participants may take:

  * Antidepressants lacking significant anticholinergic side effects
  * Estrogen replacement therapy
  * Gingko biloba is permissible, but discouraged
  * Washout from psychoactive medication (e.g., excluded antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics, etc.) for at least 4 weeks prior to screening
  * Cholinesterase inhibitors and memantine are allowable if stable for 12 weeks prior to screening

Specific Inclusion Criteria for AD participants:

* Participant must have a subjective memory concern as reported by participant, study partner, or clinician
* Abnormal memory function score on Wechsler Memory Scale (adjusted for education)
* Mini-Mental State Exam (MMSE) score between 20 and 26 (inclusive)
* Clinical Dementia Rating (CDR) = 0.5 or 1.0
* National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for probable AD
* Stability of Permitted Medications for 4 weeks. In particular, participants may take:

  * Antidepressants lacking significant anticholinergic side effects
  * Estrogen replacement therapy
  * Gingko biloba is permissible, but discouraged
  * Washout from psychoactive medication (e.g., excluded antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics, etc.) for at least 4 weeks prior to screening
  * Cholinesterase inhibitors and memantine are allowable if stable for 12 weeks prior to screening

Specific Inclusion Criteria for follow-up participants from ADNI1 and ADNI GO:

* Must have been enrolled and followed in ADNI1 for at least one year or enrolled in ADNI-GO with original diagnosis of Cognitively Normal (CN), Mild Cognitive Impairment (MCI), or Early Mild Cognitive Impairment (EMCI) regardless of whether a diagnostic conversion has occurred since initial enrollment in ADNI.
* Willing and able to continue to participate in an ongoing longitudinal study. A reduced battery of tests is allowable if the participant is not able/willing to complete the full battery.
* Study partner is available who has frequent contact with the participant (e.g. an average of 10 hours per week or more), and can accompany the participant to all clinic visits for the duration of the protocol.

Exclusion Criteria:

General (applies to each category):

* Screening/baseline MRI scan with evidence of infection, infarction, or other focal lesions; Participants with multiple lacunes or lacunes in a critical memory structure are excluded
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body
* Major depression, bipolar disorder as described in Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) within the past 1 year
* Currently treated with medication for obsessive-compulsive disorder or attention deficit disorder
* History of schizophrenia
* History of alcohol or substance abuse or dependence within the past 2 years
* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol
* Clinically significant abnormalities in B12, or TFTs that might interfere with the study
* Residence in skilled nursing facility
* Current use of specific psychoactive medications (e.g.,certain antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics, etc.); Current use of warfarin or dabigatran (exclusionary for lumbar puncture).
* Use of investigational agents one month prior to entry and for the duration of the trial
* Participation in clinical studies involving neuropsychological measures being collected more than one time per year
* Exclusion for FDG PET scan and amyloid imaging with Florbetapir F 18: Current or recent participation in any procedures involving radioactive agents such that the total radiation dose exposure to the participant in any given year would exceed the limits of annual and total dose commitment set forth in the US Code of Federal Regulations (CFR) Title 21 Section 361.1.
* Exceptions to these guidelines may be considered on a case-by-case basis at the discretion of the protocol director

Specific Exclusion Criteria for normal controls and SMC participants:

* Any significant neurologic disease, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities

Specific Exclusion Criteria for EMCI and LMCI participants:

* Any significant neurologic disease other than suspected incipient Alzheimer's disease, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.

Specific Exclusion Criteria for AD participants:

* Any significant neurologic disease other than Alzheimer's disease, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.

Specific Exclusion Criteria for follow-up participants from ADNI1 and ADNI GO:

* Participants will not be able to participate in FDG PET scan and amyloid imaging with Florbetapir F 18 if the following is true: Current or recent participation in any procedures involving radioactive agents such that the total radiation dose exposure to the participant in any given year would exceed the limits of annual and total dose commitment set forth in the US Code of Federal Regulations (CFR) Title 21 Section 361.1.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Probability Sample
Enrollment: 1182 (Actual)
Dates: Start 2011-02-14 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Rate of volume change of whole brain, hippocampus and other structural MRI measures | 5 Years

SECONDARY OUTCOMES:
Rate of Decline as measured by: Cognitive Tests, Activities of Daily Living, and CDR Sum of Boxes | 5 Years
Rate of conversion will be evaluated among all five groups | 5 Years
Rates of change on each specified biochemical biomarker | 5 Years
Rates of change of glucose metabolism (FDG-PET) | 5 Years
Extent of amyloid deposition as measured by Florbetapir F 18 | 4 Years
Group differences for each imaging and biomarker measurement | 5 Years
Correlations among biomarkers and biomarker change | 4 Years
APOE genotype, low CSF Aβ42, positive amyloid imaging with florbetapir F 18 (AV-45) | 5 Years
Rate of change of tau and extent of tau deposition as measured by flortaucipir (18F-AV-1451) | 1 Year
Rate of cognitive decline using computer based testing as measured by Cogstate Brief Battery (CBB) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Petersen, MD, PhD, Principal Investigator — Mayo Clinic; Michael W. Weiner, MD, Principal Investigator — University of California, San Francisco; Paul S. Aisen, MD, Principal Investigator — University of Southern California
Locations (58):
- United States (53):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of California, Irvine, Irvine, California
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Davis, Martinez, California
  - University of California, Irvine (Brain Imaging Center), Orange, California
  - Stanford University / PAIRE, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Wien Center for Clinical Research, Miami Beach, Florida
  - USF Health Byrd Alzheimer's Institute, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University, St. Louis, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Dartmouth Medical Center, Lebanon, New Hampshire
  - Albany Medical College, Albany, New York
  - Dent Neurologic Institute, Amherst, New York
  - New York University Medical Center, New York, New York
  - Columbia University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Beachwood, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital Memory and Aging Program, Providence, Rhode Island
  - Roper St. Francis Healthcare, North Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
- Canada (5):
  - University of British Columbia, Clinic for Alzheimer's Disease and Related Disorders Program, Vancouver, British Columbia
  - Parkwood Institute, London, Ontario
  - St. Joseph's Health Center - Cognitive Neurology, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University / Jewish General Hospital Memory Clinic, Montreal, Quebec

REFERENCES:
- [Background] Shen L, Kim S, Risacher SL, Nho K, Swaminathan S, West JD, Foroud T, Pankratz N, Moore JH, Sloan CD, Huentelman MJ, Craig DW, Dechairo BM, Potkin SG, Jack CR Jr, Weiner MW, Saykin AJ; Alzheimer's Disease Neuroimaging Initiative. Whole genome association study of brain-wide imaging phenotypes for identifying quantitative trait loci in MCI and AD: A study of the ADNI cohort. Neuroimage. 2010 Nov 15;53(3):1051-63. doi: 10.1016/j.neuroimage.2010.01.042. Epub 2010 Jan 25. PMID 20100581
- [Background] Risacher SL, Saykin AJ, West JD, Shen L, Firpi HA, McDonald BC; Alzheimer's Disease Neuroimaging Initiative (ADNI). Baseline MRI predictors of conversion from MCI to probable AD in the ADNI cohort. Curr Alzheimer Res. 2009 Aug;6(4):347-61. doi: 10.2174/156720509788929273. PMID 19689234
- [Background] Petersen RC, Aisen PS, Beckett LA, Donohue MC, Gamst AC, Harvey DJ, Jack CR Jr, Jagust WJ, Shaw LM, Toga AW, Trojanowski JQ, Weiner MW. Alzheimer's Disease Neuroimaging Initiative (ADNI): clinical characterization. Neurology. 2010 Jan 19;74(3):201-9. doi: 10.1212/WNL.0b013e3181cb3e25. Epub 2009 Dec 30. PMID 20042704
- [Background] Misra C, Fan Y, Davatzikos C. Baseline and longitudinal patterns of brain atrophy in MCI patients, and their use in prediction of short-term conversion to AD: results from ADNI. Neuroimage. 2009 Feb 15;44(4):1415-22. doi: 10.1016/j.neuroimage.2008.10.031. Epub 2008 Nov 5. PMID 19027862
- [Derived] Miller AA, Sharp ES, Wang S, Zhao Y, Mecca AP, van Dyck CH, O'Dell RS; Alzheimer's Disease Neuroimaging Initiative (ADNI). Self-reported hearing loss is associated with faster cognitive and functional decline but not diagnostic conversion in the ADNI cohort. Alzheimers Dement. 2024 Nov;20(11):7847-7858. doi: 10.1002/alz.14252. Epub 2024 Sep 26. PMID 39324520
- [Derived] Howe MD, Caruso MR, Manoochehri M, Kunicki ZJ, Emrani S, Rudolph JL, Huey ED, Salloway SP, Oh H; Alzheimer's Disease Neuroimaging Initiative. Utility of cerebrovascular imaging biomarkers to detect cerebral amyloidosis. Alzheimers Dement. 2024 Oct;20(10):7220-7231. doi: 10.1002/alz.14207. Epub 2024 Sep 1. PMID 39219209
- [Derived] Howe MD, Caruso MR, Manoochehri M, Kunicki ZJ, Emrani S, Rudolph JL, Huey ED, Salloway SP, Oh H; Alzheimer's Disease Neuroimaging Initiative. Utility of cerebrovascular imaging biomarkers to detect cerebral amyloidosis. medRxiv [Preprint]. 2024 May 28:2024.05.28.24308056. doi: 10.1101/2024.05.28.24308056. PMID 38853879
- [Derived] Rauchmann BS, Schneider-Axmann T, Perneczky R; Alzheimer's Disease Neuroimaging Initiative (ADNI). Associations of longitudinal plasma p-tau181 and NfL with tau-PET, Abeta-PET and cognition. J Neurol Neurosurg Psychiatry. 2021 Dec;92(12):1289-1295. doi: 10.1136/jnnp-2020-325537. Epub 2021 Jun 29. PMID 34187867
- See also: Alzheimer's Therapeutic Research Institute — https://keck.usc.edu/atri/
- See also: Laboratory of Neuroimaging: Alzheimer's Disease Neuroimaging Initiative — http://adni.loni.usc.edu/
- See also: Alzheimer's Disease Neuroimaging Initiative — http://adni.loni.usc.edu/
- See also: List of Alzheimer's Disease Neuroimaging Initiative Publications — http://adni.loni.usc.edu/news-publications/publications/